CLINICAL TRIAL: NCT04676464
Title: VALIDation of Bedside Ultrasound of Muscle Layer Thickness of the Quadriceps in the Critically Ill Patient: The VALIDUM Study
Brief Title: VALIDation of Bedside Ultrasound of Muscle Layer Thickness of the Quadriceps in the Critically Ill Patient
Acronym: VALIDUM
Status: Completed | Type: Observational
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Director of Clinical Evaluation Research Unit, Queen's University
Other Study IDs: VALIDUM
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness; Muscle Atrophy
Keywords: computed tomography; muscle atrophy; muscle thickness; intensive care unit; ultrasound
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultra- sound: ultra- sound assessment of their quadriceps muscle layer thickness (QMLT)
  Interventions: Diagnostic Test: Ultra- sound

INTERVENTIONS:
Diagnostic Test: Ultra- sound — Ultrasound assessment of quadricep muscle layer thickness QMLT within 72hrs of initial CT scan

SUMMARY:
The overall objective is to evaluate the validity of bedside US of QMLT and MF-BIA by comparing measurements from US and MF-BIA to those estimates of lean body mass obtained from CT Scan of abdomen when done for clinical reasons.

The investigators expect to observe a high degree of correlation between these 3 baseline measures and the changes in US measures and MF-BIA over time to correlate with changes to CT Scan measures of lean body mass.

DETAILED DESCRIPTION:
The overall objective is to evaluate the validity of bedside US of QMLT and MF-BIA by comparing measurements from US and MF-BIA to those estimates of lean body mass obtained from CT Scan of abdomen when done for clinical reasons.

The investigators expect to observe a high degree of correlation between these 3 baseline measures and the changes in US measures and MF-BIA over time to correlate with changes to CT Scan measures of lean body mass.

This is a multi center, prospective, observation study across 5-6 intensive care units which will enroll 200 participants over a 12 month enrollment period followed by a 6 month period to complete data analysis.

This study will enroll a broad heterogeneous participant population who will be admitted to the ICU for inpatient care. We are particularly interested in the cohort of participant with trauma but will enroll non-trauma participants who have CT scans as well to do some between group comparisons. Participants enrolled to this study will be followed until they are discharged from the index hospital.

This is a prospective, observational study therefore no specific interventions will be associated with this study. The following information will be collected and recorded during ICU and hospital stay:

CT Images - All abdominal CT images conducted during the index hospitalization ordered for clinical purposes will be retrieved to precisely quantify muscle and adipose tissue mass.

Ultrasound - A portable ultrasound will be completed as soon as possible following the initial CT Scan, and again while a participant remains in hospital for each follow up CT of the abdomen for clinical reasons, where feasible, unless it is within a week of the previous CT scan.

Multiple Frequency Bioelectrical Impedance Analysis (MF-BIA) -MF-BIA is a non-invasive and simple-to-use method of measuring body composition and nutritional status in the clinical setting. MF-BIA measurements will be conducted every time an US measurement is done in the ICU following a CT Scan done for clinical reasons, unless it is within a week of the previous CT Scan and accompanying MF-BIA. After discharge from the ICU to the hospital, where feasible, MF BIA will be done every time an ultrasound is done following CT scans done for clinical reasons, unless it is within a week of the previous CT Scan and accompanying MF-BIA. MF-BIA will not be done on individuals with a pacemaker, Baseline patient demographics data and nutritional adequacy data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal CT scan performed for clinical reasons within 24 hours before or 72 hours after admission

Exclusion Criteria:

* Patients under age 18 years
* Moribund patient with devastating injuries and not expected to survive
* Patients whose clinical condition precludes performing an ultrasound
* Pregnant women
* Prisoners
* Mentally-disabled individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll a broad heterogeneous patient population who will be admitted to the ICU for inpatient care. We are particularly interested in the cohort of patients with trauma but will enroll non-trauma patients who have CT scans as well to do some between group comparisons.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validity of bedside US of QMLT | 12 months
  To evaluate the validity and reliability of bedside US by comparing measurements from US and to those estimates of lean body mass obtained from CT Scan of abdomen.

IPD SHARING:
Plan to Share IPD: No